CLINICAL TRIAL: NCT05424913
Title: Exploratory Study of the Relationships Between the Biomarkers of Inflammation, Lipidome and Insulin Resistance and Disorders of Glycemic Regulation in a Cohort of Insulin-resistant Subjects Due to Excess Weight or Dunnigan's Lipodystrophy
Acronym: IRAP-DUN 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2017/CHU/07-2021-A00105-36
Record Dates: First submitted 2022-06-03; First posted 2022-06-21 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2022-06

CONDITIONS: Lipodystrophy; Dunnigan Syndrome
MeSH Terms: conditions — Lipodystrophy; Lipodystrophy, Familial Partial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Subjects with Dunnigan's Lipodystrophy (Other)
  Interventions: Other: research-specific blood sample
- Non-lipodystrophic insulin-resistant subjects (Other)
  Interventions: Other: research-specific blood sample
- Insulin-sensitive non-lipodystrophic subjects (Other)
  Interventions: Other: research-specific blood sample

INTERVENTIONS:
Other: research-specific blood sample — blood sample of 50 ml maximum levels of serum Insulin Regulated Amino Peptidase, lipidome markers and inflammation markers

SUMMARY:
The objective of this work is to identify biomarkers of interest in patients with insulin resistance leading to early disorders of glycemic regulation. For this the investigators want to assay the insulin resistance marker Insulin Regulated Amino Peptidase serique (IRAPs), the plasma lipidome and inflammation markers in 2 populations of insulin-resistant subjects due to Dunnigan's inherited lipodystrophy or overweight/obesity and insulin-sensitive subjects with or without a glycemic regulation disorder objectified during an Oral induced hyperglycemia. The results of the IRAPs, lipidome and inflammation assays will be compared in insulin-resistant subjects, between normoglycemic, prediabetic and diabetic subjects. Correlations will be made between these markers and the deterioration of glycemic regulation as well as with known insulin resistance parameters (HOmeostasis Assessment Model (HOMA), Quantitative Insulin-sensitivity Check Index (QUICKI),Insulin Sensitivity Index (Isi) MATSUDA).

ELIGIBILITY:
Inclusion Criteria:

* Subjects with Dunnigan's Lipodystrophy OR Non-lipodystrophic insulin-resistant subjects OR Insulin-sensitive non-lipodystrophic subjects
* major
* Subjects benefiting from metabolic exploration in the Endocrinology, Diabetology and Nutrition department of the Reunion University Hospital.
* Subject benefiting from an oral glucose tolerance test (OGTT) during his follow-up in the Endocrinology, Diabetology and Nutrition department of the Reunion University Hospital.
* Person affiliated or beneficiary of a social security scheme.
* Subject having been informed of the study in progress and having given their written consent.

Exclusion Criteria:

* Pregnant woman
* Person under guardianship or curators or deprived of liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2021-08-17 (Actual); Primary Completion 2023-08-16 (Actual); Study Completion 2023-08-16 (Actual)

PRIMARY OUTCOMES:
Insulin Regulated Amino Peptidase sérique (IRAPs) levels | at inclusion
  Insulin Regulated Amino Peptidase sérique (IRAPs)
inflammation markers levels | at inclusion
  TNF-α (tumor necrosis factors-α), IL-1β (interleukin-1β), IL-2, IL-6, IL-18, IFN-γ (interferon-γ) et MCP-1 (monocyte chemoattractant protein-1), IL-10, IL-4, IL-5
lipidome markers levels | at inclusion
  662 plasma lipid species

SECONDARY OUTCOMES:
Compare levels of Insulin Regulated Amino Peptidase sérique (IRAPs) between the 3 categories of participants | at inclusion
  Insulin Regulated Amino Peptidase sérique (IRAPs)
Compare levels of inflammation markers between the 3 categories of participants | at inclusion
  TNF-α (tumor necrosis factors-α), IL-1β (interleukin-1β), IL-2, IL-6, IL-18, IFN-γ (interferon-γ) et MCP-1 (monocyte chemoattractant protein-1), IL-10, IL-4, IL-5
Compare levels of lipidome markers between the 3 categories of participants | at inclusion
  662 plasma lipid species

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de la Réunion, Saint-Pierre, Reunion

IPD SHARING:
Plan to Share IPD: No